CLINICAL TRIAL: NCT02578225
Title: Acute and Chronic Heart Failure in Real Life in Turkey: National, Multi-center, Epidemiological, Observational and Ad-Hoc Cross-sectional Study
Brief Title: Snapshot Evaluation of Acute and Chronic Heart Failure in Real Life in Turkey
Acronym: SELFIE-TR
Status: Completed | Type: Observational
Sponsor: Prof. Dr. Mehmet Birhan Yılmaz (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Mehmet Birhan Yılmaz, Prof. Dr., Cumhuriyet University
Organization: Cumhuriyet University (Other)
Other Study IDs: 288-AU/003
Record Dates: First submitted 2015-08-28; First posted 2015-10-16 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Chronic Heart Failure
Keywords: Heart; Chronic; Failure; MI; real life; Turkey
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Non interventional study

SUMMARY:
This study, which will be conducted at 23 sites representing the determined NUTS-1 regions in Turkey, in which all patients who were admitted to clinic or were hospitalized with Heart Failure (Acute or Chronic) diagnosis will be enrolled into the study, for a month and on a day of the week which will be determined by the site itself, is a national, multi-center, observational, epidemiological and cross-sectional study. This study is a local study which is planned to be conducted only in Turkey. Included patients of the study will be clinically evaluated by the physicians who are maintaining them and will receive the standard medical treatment which is determined by their physicians in normal life conditions. No experimental intervention or treatment will be received by patients in relation to the enrollment to this study. Therefore, this study does not contain a protocol or a pre-determined visit flowchart. However, patients with Heart Failure diagnosis should grant their consent to the retrospective utilization of their data and questions which will be asked to them about their disease history. Provided that the study's design is non-pharmacological observational, investigators will treat and follow the patients in accordance with their own medical decisions and their best clinical experiences.

"Snapshot Evaluation of Heart Failure in Turkey: Initial Analysis from SELFIE-TR"

DETAILED DESCRIPTION:
STUDY DESIGN STEPS

1. The steps described below will be taken in accordance with ICD code for acute and chronic heart failure patients with a verified heart failure diagnosis:

* Verification of patient's heart failure diagnosis according to ICD code.
* In order to include the patient to the study, signing of the consent form.
* Documentation of patient demographics, medical history, heart failure history, co-morbidities and risk factors.
* Prospective recording of findings of physical examination.
* Retrospective recording of results related to diagnostic methods (biochemistry, blood count and others).
* Determination of NYHA classification.
* Determination of pathophysiology and etiology.
* Recording treatment patterns.
* Inspection of patient's device usage status (pacemaker, ICD, CRT, LVAD, transplantation).
* Inspection of hospitalization rates.

SELFIE-HF study starting date is planned as month September of 2015 and it is planned that the physicians will execute study enrollment on an allocated day of the week for 4 weeks. It is also planned that the data collected on months October and November will be inspected and listed and patients will be contacted by phone after 1 year after enrolment date in order to inquire about survival status. Therefore, estimated termination date of the study, with patient follow-up calls, is planned to be the last quarter of 2016.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and older male and female patients
* Disregarding the consultation method or the severity of disease, Acute Heart Failure patients who have been hospitalized
* Chronic Heart Failure patients who have been admitted to clinic
* Patients who have agreed to participate to the study

Exclusion Criteria:

* Patients who have expressed their rejection for study participation
* Patients without a Heart Failure Diagnosis or whose diagnosis is changed or deemed uncertain during index application

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In 23 designated sites, for a month on a day which will be determined by the site itself, patients who have been admitted to the clinic or hospitalized with Heart Failure (Acute and Chronic) diagnosis will be enrolled into the study. Target population of the study is the acute and chronic heart failure patients who will consult to the hospital on the related day of the week for a month which is determined by sites.
Sampling Method: Probability Sample
Enrollment: 1054 (Actual)
Dates: Start 2015-10; Primary Completion 2016-09 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Survival in patients with acute and chronic heart failure | >1 year after the enrollment is over
  Patients with acute and chronic heart failure will be contacted via telephone call at least 1 year after the enrollment to see their survival status and cardiovascular mortality rates will be calculated as an outcome measure and will be compared (acute versus chronic).

SECONDARY OUTCOMES:
Guideline directed heart failure medications and outcome | Prospective data collection during follow up
  Prescription records of patients will be obtained and patients will be classified into two as those with and those without specific prescribed medication, and then these findings will be related to cardiovascular mortality
Co-morbidities and outcome | Prospective survival data collection during follow up
  Records of patients with regard to existing co-morbidities during index event will be collected and then be related to cardiovascular mortality during follow up.

CONTACTS AND LOCATIONS:
Locations (23):
- Turkey (Türkiye) (23):
  - Cukurova University School of Medicine, Adana
  - Kocatepe University School of Medicine, Afyonkarahisar
  - Hacettepe University School of Medicine, Ankara
  - Yüksek İhtisas Training and Research Hospital, Ankara
  - Adnan Menderes University School of Medicine, Aydin
  - Hitit University School of Medicine, Çorum
  - Trakya University School of Medicine, Edirne
  - Firat University School of Medicine, Elâzığ
  - Ataturk University School of Medicine, Erzurum
  - İstanbul University Cardiology Institute, Istanbul
  - Siyami Ersek Training and Research Hospital, Istanbul
  - Ege University School of Medicine, Izmir
  - İzmir Tepecik Training And Research Hospital, Izmir
  - Kilis State Hospital, Kilis
  - Kocaeli University School of Medicine, Kocaeli
  - Kirikkale University School of Medicine, Kırıkkale
  - Inonu University School of Medicine, Malatya
  - Sutcu Imam University School of Medicine, Maras
  - Mersin University School of Medicine, Mersin
  - Sakarya University School of Medicine, Sakarya
  - Ondokuz Mayis University School of Medicine, Samsun
  - Cumhuriyet University School of Medicine, Sivas
  - Karadeniz Technical University School of Medicine, Trabzon